CLINICAL TRIAL: NCT01882426
Title: A Cluster Randomized Controlled Trial of a Care-Path for the Management of Ulcerative Colitis
Brief Title: Care Path for the Management of Ulcerative Colitis
Acronym: CONSTRUCT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP1206
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Ulcerative Colitis
Keywords: CONSTRUCT; Cluster randomization controlled trial; Gastroenterology practices in North America
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced treatment algorithm (Active Comparator): Treatment algorithm featuring the early use of combination therapy, treatment intensification guided by objective assessments of inflammation and the use of remission as a therapeutic goal
  Interventions: Other: Enhanced treatment algorithm
- Usual Care (Placebo Comparator): These subjects will be managed according to local treatment guidelines for the treatment of UC.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Enhanced treatment algorithm — Practitioners assigned to the intervention arm will be educated on the use of the Enhanced Algorithm.
  Arms: Enhanced treatment algorithm
Other: Usual Care — usual step care practice
  Arms: Usual Care

SUMMARY:
Assess if standardized care-path that features objective evaluations of disease activity and time-bound algorithms is superior to usual step-care in the treatment of ulcerative colitis.

DETAILED DESCRIPTION:
Step-care based on symptomatic response remains the overwhelming algorithm of choice in clinical practice. Many subjects receive infliximab only as a last resort, when the subject is very ill and has failed repeated attempts of corticosteroid induction therapy. Although this situation is far from ideal, to change such entrenched physician behavior will require compelling evidence that Step-care results in inferior outcomes to earlier introduction of effective therapy.

Based on these considerations, we will perform a cluster randomization trial in which 40 gastroenterology practices will be randomly assigned to a treatment algorithm featuring the early use of combination therapy, treatment intensification guided by objective assessments of inflammation and the use of remission as a therapeutic goal or a conventional Step-care approach.

ELIGIBILITY:
Inclusion Criteria:

* Females of child bearing potential must have a negative serum pregnancy test prior to randomization, and must use a hormonal (oral, implantable or injectable) or barrier method of birth control throughout the study. Females unable to bear children must have documentation of such in the source records -- - Documented diagnosis of UC with a Mayo Clinic Score (MCS) ≥6 and a baseline Mayo Endoscopy Score >2.
* Either an elevated serum C-reactive protein (CRP) (above the Upper Level of Normal (ULN) according to local laboratory results) or elevated fecal calprotectin (> 250 mg/kg) concentration.
* Requires sigmoidoscopic evaluation at baseline (standard of care)
* Written informed consent must be obtained and documented.
* Ability of subject to participate fully in all aspects of this clinical trial in the opinion of the investigator.

Exclusion Criteria:

* Previous failure of TNF antagonist therapy
* Received any investigational drug in the past 30 days or 5 half-lives, whichever is longer.
* Pregnant or lactating women.
* Any conditions (e.g., history of alcohol or substance abuse) which in the opinion of the investigator, may interfere with the subject's ability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in remission at the end of 12 months. | 12 months
  Remission is defined as 1) a Mayo Clinic Score of ≤2 with rectal bleeding and stool frequency sub-scale scores of 0) with no use of corticosteroids, and 3) normalization of the subject's index inflammatory marker (c-reactive protein or calprotectin). The primary endpoint will be assessed at Month 12.

SECONDARY OUTCOMES:
Proportion of patients in remission over the course of the study | 18 months
  The time in remission over the course of the study; occurrence of surgery or hospitalization for Ulcerative Colitis; occurrence of disease-related complications; health related QoL (Short-Form 36 questionnaire [SF-36] and EuroQoL instrument [EQ-5D]); and, subject

CONTACTS AND LOCATIONS:
Overall Officials: Brian G Feagan, MD, Principal Investigator — Alimentiv Inc.

REFERENCES:
- [Background] Kornbluth A, Sachar DB; Practice Parameters Committee of the American College of Gastroenterology. Ulcerative colitis practice guidelines in adults: American College Of Gastroenterology, Practice Parameters Committee. Am J Gastroenterol. 2010 Mar;105(3):501-23; quiz 524. doi: 10.1038/ajg.2009.727. Epub 2010 Jan 12. PMID 20068560
- [Background] D'Haens G, Baert F, van Assche G, Caenepeel P, Vergauwe P, Tuynman H, De Vos M, van Deventer S, Stitt L, Donner A, Vermeire S, Van De Mierop FJ, Coche JR, van der Woude J, Ochsenkuhn T, van Bodegraven AA, Van Hootegem PP, Lambrecht GL, Mana F, Rutgeerts P, Feagan BG, Hommes D; Belgian Inflammatory Bowel Disease Research Group; North-Holland Gut Club. Early combined immunosuppression or conventional management in patients with newly diagnosed Crohn's disease: an open randomised trial. Lancet. 2008 Feb 23;371(9613):660-667. doi: 10.1016/S0140-6736(08)60304-9. PMID 18295023
- [Background] Colombel JF, Sandborn WJ, Reinisch W, Mantzaris GJ, Kornbluth A, Rachmilewitz D, Lichtiger S, D'Haens G, Diamond RH, Broussard DL, Tang KL, van der Woude CJ, Rutgeerts P; SONIC Study Group. Infliximab, azathioprine, or combination therapy for Crohn's disease. N Engl J Med. 2010 Apr 15;362(15):1383-95. doi: 10.1056/NEJMoa0904492. PMID 20393175
- [Background] Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med. 1987 Dec 24;317(26):1625-9. doi: 10.1056/NEJM198712243172603. PMID 3317057
- [Background] D'Haens G, Sandborn WJ, Feagan BG, Geboes K, Hanauer SB, Irvine EJ, Lemann M, Marteau P, Rutgeerts P, Scholmerich J, Sutherland LR. A review of activity indices and efficacy end points for clinical trials of medical therapy in adults with ulcerative colitis. Gastroenterology. 2007 Feb;132(2):763-86. doi: 10.1053/j.gastro.2006.12.038. Epub 2006 Dec 20. No abstract available. PMID 17258735